CLINICAL TRIAL: NCT06905171
Title: Analysis of Brain Responses and Habituation to Multimodal Sensory Stimuli in Patients With Fibromyalgia
Brief Title: Habituation of Brain Responses to Sensory Stimuli in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, José Biurrun Manresa, PhD, National Council of Scientific and Technical Research, Argentina
Other Study IDs: IS004760
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
Keywords: Event-Related Potentials; Electroencephalography; Habituation
MeSH Terms: conditions — Fibromyalgia; Substance-Related Disorders | interventions — Acoustic Stimulation; Photic Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fibromyalgia Patients: Patients with primary fibromyalgia diagnosis. May include other chronic pain comorbidities, but the pain associated with those diseases should be less severe than the pain caused by fibromyalgia.
  Interventions: Other: Auditory Stimulation; Other: Visual Stimulation; Other: Somatosensory Stimulation; Other: Auditory-Visual Stimulation; Other: Visual-Somatosensory Stimulation; Other: Auditory-Somatonsensory Stimulation; Other: Auditory-Visual-Somatosensory Stimulation
- Healthy Controls: Volunteers with no clinical history of chronic pain, musculoskeletal or articular disorders
  Interventions: Other: Auditory Stimulation; Other: Visual Stimulation; Other: Somatosensory Stimulation; Other: Auditory-Visual Stimulation; Other: Visual-Somatosensory Stimulation; Other: Auditory-Somatonsensory Stimulation; Other: Auditory-Visual-Somatosensory Stimulation

INTERVENTIONS:
Other: Auditory Stimulation — A tone at a 1000 Hz frequency, delivered through speakers at a comfortable volume
Other: Visual Stimulation — A checkerboard pattern displayed on a monitor, with colors alternating every 25 ms
Other: Somatosensory Stimulation — A train of three electrical stimuli, each lasting 1 ms, separated by 8 ms, at an intensity that clearly elicits a pricking sensation
Other: Auditory-Visual Stimulation — Stimulation using auditory and visual stimuli concomitantly
Other: Visual-Somatosensory Stimulation — Stimulation using visual and somatosensory stimuli concomitantly
Other: Auditory-Somatonsensory Stimulation — Stimulation using auditory and somatosensory stimuli concomitantly
Other: Auditory-Visual-Somatosensory Stimulation — Stimulation using auditory, visual and somatosensory stimuli concomitantly

SUMMARY:
The goal of this observational study is to assess event-related potentials and habituation in patients with fibromyalgia. The main research questions are:

* Is there a measurable difference in sensory responses between fibromyalgia patients and healthy control?
* Could these measures provide evidence supporting claims of hypersensitivity?

Participants will:

- receive randomized sensory stimuli (auditory, visual, somatosensory, audiovisual, auditory-somatosensory, visual-somatosensory, and auditory-visual-somatosensory) in blocks of 20 trials.

DETAILED DESCRIPTION:
Fibromyalgia is a disorder characterized primarily by widespread musculoskeletal pain. It is often accompanied by symptoms such as fatigue, insomnia, cognitive difficulties, etc. In addition to chronic pain, patients frequently report hypersensitivity to sensory stimuli, both nociceptive and non-nociceptive. Studies using psychophysical and electrophysiological tests have found altered sensory processing in fibromyalgia patients.

Research focused on event-related potentials (ERPs) have found differences in amplitude in the responses to auditory, nociceptive, and non-nociceptive somatosensory stimuli in fibromyalgia patients . One key aspect evaluated through ERPs is habituation, defined as a decrease in response due to repeated stimulation. In healthy individuals, ERPs amplitude decreases with repeated sensory input due to progressive neuronal response reduction. In fibromyalgia patients, reduced habituation has been observed for laser-induced ERPs and somatosensory ERPs, though no differences were found for auditory ERPs.

ERPs not only provide information about sensory modalities but also contain non-specific components related to stimulus expectation, motor preparation, and attentional orientation. Previous studies have attempted to isolate this non-specific component, as part of habituation may stem from a decrease in its amplitude rather than from a direct sensory response reduction. Using an analytical model, researchers successfully separated this component in experiments with individually or simultaneously presented stimuli, yielding promising results.

In the present study, participants (both fibromyalgia patients and healthy controls) will attend one experimental session in which stimulation in different sensory modalities will take place along with electroencephalographic (EEG) recordings. For each stimulus type, 2 blocks of 20 trials will be performed.The order of the stimulus will be selected randomly, but they can be divided into three categories:

* Unimodal stimulus

  * Auditory (A): a 1000 Hz tone delivered at a comfortable volume through a speaker
  * Visual (V): a checkerboard pattern, inverted every 25 ms, presented on a computer screen.
  * Somatosensory (S): a train of 3 electrical stimuli that elicits a pricking sensation.
* Bimodal stimulus

  * Auditory-Visual (AV)
  * Auditivo-Somatosensory (AS)
  * Visual-Somatosensory (VS)
* Trimodal Stimulus

  * Auditory-Visual-Somatosensory (AVS) The aim of the study is to evaluate neurophysiological parameters related to habituation in multimodal sensory stimulation environments to characterize ERPs in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

Fibromyalgia patients:

* Primary diagnosis of fibromyalgia according to the criteria used by the healthcare professional in charge of the patient.
* Other comorbidities are accepted as long as the pain caused by them is less severe than the pain caused by fibromyalgia.
* Willingness and ability to fully understand the content and scope of the experiment and to comply with the experiment instructions.
* Normal or corrected-to-normal vision.
* Normal hearing

Healthy controls:

* No history of neurological diseases, chronic pain or musculoskeletal disorders.
* Willingness and ability to fully understand the content and scope of the experiment and to comply with the experiment instructions.
* Normal or corrected-to-normal vision.
* Normal hearing

Exclusion Criteria:

Fibromyalgia patients:

* Pregnancy
* History of addictive behavior, defined as alcohol, cannabis, opioids or other drugs abuse.
* Presence of fever, tuberculosis, malignant tumors, infectious processes, acute inflammatory processes.
* Lack of cooperation

Healthy controls:

* Pregnancy
* History of chronic pain or musculoskeletal or articular disorders
* History of addictive behavior, defined as alcohol, cannabis, opioids or other drugs abuse.
* Presence of fever, tuberculosis, malignant tumors, infectious processes, acute inflammatory processes.
* Lack of cooperation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohorts of patients and healthy controls wil be selected from the city of Paraná and surrounding areas. Through the ONG "Fibromialgia Entre Ríos Asociación Civil", the patients will be reached out and asked wether or not they are willing to participate. Additionally, flyer will be hung in major health facilities in the city and made public on social media. The cohort of healthy volunteers will be recruited after the patients for age, genre and socieconomic matching
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Percentual Habituation | Immediately after the intervention
  Relative reduction in the amplitude of evoked potentials between consecutive stimuli

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire-Revised version (FIQR) | 10 minutes before the intervention
  Instrument for the assessment and evaluation of fibromyalgia patient's status. Scores range from 0 to 100, with a higher number indicating more impacts of fibromyalgia symptoms in daily life
Symptoms Impact Questionnaire (SIQ) | 10 minutes before the intervention
  Instrument to assess healthy control's status regarding relevant clinical symptoms experienced in the last week. Scores range from 0 to 100, with a higher number indicating more impacts of their symptoms in daily life activities
Hospital Anxiety and Depression Scale (HADS) | 10 minutes before the intervention
  Widely used instrument to evaluate anxiety and depression. It is divided into 7 questions assessing anxiety and 7 assessing depression. The scores range from 0 to 21, with higher scores indicating worse clinical symptoms.
Numeric Rating Scale Pain (NRSp) | 10 minutes before the intervention
  Pain at the moment of the experimental session. Scores range from 0 to 10, with higher number indicating worse pain.
Stimulus saliency | Immediately after the intervention
  A number reflecting the ability of a stimulus to stand out relative to the sensory background or relative to the preceding stimuli
Event-related potentials amplitude | Immediately after the intervention
  Amplitude, in microvolts, of event-related brain potentials
Event-related potentials latency | Immediately after the intervention
  Latency, in milliseconds, of event-related brain potentials
Non-specific components amplitude | Immediately after the intervention
  Amplitude, in microvolts, of the non/specific component derived from the ERPs
Non-specific components latency | Immediately after the intervention
  Latency, in milliseconds, of the non-specific component derived from the ERPs

CONTACTS AND LOCATIONS:
Overall Officials: Biurrun Manresa, Principal Investigator — National Council of Scientific and Technical Research, Argentina (CONICET)
Locations (1):
- Faculty of Engineering-National University of Entre Ríos, Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available on the 'Open Science Framework' after undergoing the process of anonymization to remove any participant-identifying information. The data will consist of the raw EEG signals and raw behavioral responses to cognitive tasks. Additionally, the statistical analysis and Jupyter notebooks used to process the data will also be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The participant's data and the processing pipeline will be available after the data collection is finished. The supporting information (including the study protocol, the statistical analysis plan and the informed consent) will be uploaded as soon as possible.
Access Criteria: The data will be publicly available.

REFERENCES:
- [Background] Gondan M, Roder B. A new method for detecting interactions between the senses in event-related potentials. Brain Res. 2006 Feb 16;1073-1074:389-97. doi: 10.1016/j.brainres.2005.12.050. Epub 2006 Jan 20. PMID 16427613
- [Background] Thompson RF, Spencer WA. Habituation: a model phenomenon for the study of neuronal substrates of behavior. Psychol Rev. 1966 Jan;73(1):16-43. doi: 10.1037/h0022681. No abstract available. PMID 5324565
- [Background] Montoya P, Sitges C, Garcia-Herrera M, Rodriguez-Cotes A, Izquierdo R, Truyols M, Collado D. Reduced brain habituation to somatosensory stimulation in patients with fibromyalgia. Arthritis Rheum. 2006 Jun;54(6):1995-2003. doi: 10.1002/art.21910. PMID 16732548
- [Background] Lorenz J. Hyperalgesia or hypervigilance? An evoked potential approach to the study of fibromyalgia syndrome. Z Rheumatol. 1998;57 Suppl 2:19-22. doi: 10.1007/s003930050228. PMID 10025076
- [Background] de Tommaso M, Federici A, Santostasi R, Calabrese R, Vecchio E, Lapadula G, Iannone F, Lamberti P, Livrea P. Laser-evoked potentials habituation in fibromyalgia. J Pain. 2011 Jan;12(1):116-24. doi: 10.1016/j.jpain.2010.06.004. Epub 2010 Aug 4. PMID 20685171
- [Background] Alanoglu E, Ulas UH, Ozdag F, Odabasi Z, Cakci A, Vural O. Auditory event-related brain potentials in fibromyalgia syndrome. Rheumatol Int. 2005 Jun;25(5):345-9. doi: 10.1007/s00296-004-0443-3. Epub 2004 Feb 21. PMID 14986061
- [Background] McDermid AJ, Rollman GB, McCain GA. Generalized hypervigilance in fibromyalgia: evidence of perceptual amplification. Pain. 1996 Aug;66(2-3):133-44. doi: 10.1016/0304-3959(96)03059-x. PMID 8880834
- [Background] Young EL, Mista CA, Jure FA, Andersen OK, Biurrun Manresa JA. An analytical method to separate modality-specific and nonspecific sensory components of event-related potentials. Eur J Neurosci. 2022 Oct;56(7):5090-5105. doi: 10.1111/ejn.15798. Epub 2022 Aug 31. PMID 35983754
- [Background] Staud R, Godfrey MM, Robinson ME. Fibromyalgia Patients Are Not Only Hypersensitive to Painful Stimuli But Also to Acoustic Stimuli. J Pain. 2021 Aug;22(8):914-925. doi: 10.1016/j.jpain.2021.02.009. Epub 2021 Feb 23. PMID 33636370
- [Background] Lim M, Roosink M, Kim JS, Kim HW, Lee EB, Son KM, Kim HA, Chung CK. Augmented Pain Processing in Primary and Secondary Somatosensory Cortex in Fibromyalgia: A Magnetoencephalography Study Using Intra-Epidermal Electrical Stimulation. PLoS One. 2016 Mar 18;11(3):e0151776. doi: 10.1371/journal.pone.0151776. eCollection 2016. PMID 26992095